CLINICAL TRIAL: NCT01656772
Title: Vdrive Evaluation of Remote Steering and Testing in Lasso Electrophysiology Procedures Study
Acronym: VERSATILE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stereotaxis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-020
Record Dates: First submitted 2012-07-30; First posted 2012-08-03 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation
Keywords: magnetic navigation; robotic control; RMT ThermoCool catheter
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual Lasso navigation (Active Comparator): Use of conventional manual navigation techniques with the Lasso catheter
  Interventions: Procedure: Manual Lasso navigation
- Vdrive Lasso navigation (Experimental): Use of the Vdrive to remotely and robotically control the manipulation of a Lasso catheter
  Interventions: Device: Vdrive Lasso navigation

INTERVENTIONS:
Device: Vdrive Lasso navigation — Remote robotic Lasso navigation
  Arms: Vdrive Lasso navigation
Procedure: Manual Lasso navigation — Manually maneuver a Lasso catheter
  Arms: Manual Lasso navigation

SUMMARY:
This study will evaluate the use of a robotic device that is remotely controlled to maneuver a circular mapping catheter in the left atrium during Atrial Fibrillation (AF) ablation procedures.

DETAILED DESCRIPTION:
Key to the success of an electrophysiology procedure is the ability to accurately map, sense and pace the heart. Electrophysiology mapping catheters are available in a variety of shapes and electrode configurations. The majority of these catheters are manipulated manually by the physician. The Vdrive simplifies these manipulations by allowing an operator to mechanically advance, retract, rotate, deflect and maneuver a circular mapping catheter. The circular mapping catheter is not altered in structure, function or indication in the same manner as the predicate device (Cardiodrive Catheter Advancement System).

This is a prospective, randomized, non-blinded, controlled study comparing manual navigation of a circular mapping catheter with mechanical navigation by the Vdrive. A total of 120 patients are expected to complete the study: 80 patients in the Vdrive navigation arm and 40 patients in the manual navigation arm. Patients will be enrolled at a minimum of one site in the European Union where the product is currently marketed and the United States, where the Vdrive is considered to be investigational.

ELIGIBILITY:
Inclusion Criteria:

* Left atrial AF ablation procedure requiring the use of a Lasso mapping catheter
* Subject must be at least 18 years of age
* Subject must be male, female of no childbearing potential, or a female that has a negative pregnancy test prior to randomization

Exclusion Criteria:

* Unable to safely expose subject to a magnetic field
* Prior AF ablation procedure
* Patients with fewer than 4 PVs are excluded
* Patients with persistent AF in whom early recurrence of AF following cardioversion would preclude completion of the pacing maneuvers described in the protocol or patients with other conditions that would similarly preclude completion of the pacing maneuvers
* Contraindication to procedure or unable to return for follow-up
* History of clotting disorder, bleeding abnormalities or contraindication to anticoagulation
* Actively participating in other cardiac device trial(s)
* Currently pregnant
* Under 18 years of age
* Prosthetic valves
* Atrial abnormalities (thrombus, myxoma or baffle)
* Other exclusions per the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qun Sha, MD, Study Director — Stereotaxis Inc
Locations (5):
- United States (3):
  - Central Baptist Hospital, Lexington, Kentucky
  - Texas Cardiac Arrhythmia Institute, Austin, Texas
  - Baylor Research Institute, Dallas, Texas
- ZNA Campus Middelheim Lindendreef 1, Antwerp, Antwerpen, Belgium
- IKFE HDZ GbmH, Bad Oeynhausen, Bad Oeynhausen, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Manual Lasso Navigation | Vdrive Lasso Navigation
Started | 43 | 77
Completed | 43 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual Lasso Navigation | Vdrive Lasso Navigation | Total
Number analyzed (Participants) | 43 | 77 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.2) | 62.4 (9.8) | 62.6 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 34 | 63 | 97
Region of Enrollment [Number; unit: participants]
  Belgium | 11 | 23 | 34
  United States | 20 | 33 | 53
  Germany | 12 | 21 | 33

OUTCOME MEASURES:

1. Primary Outcome: The Primary Effectiveness Endpoint is the Successful Navigation and EGM Recording of Each Pre-specified Pulmonary Vein Per Procedure Between Both the Control and the Investigational Device Groups.
Description: Success was navigating and sensing by obtaining an EGM at the pre-specified targeted PVs. The null hypothesis was to be tested at the α = 0.05 significance level using a test statistic Z based on the Farrington and Manning likelihood score statistic with adjustment to take into account the correlation between multiple observations (PVs) on the same subject. The null hypothesis was to be rejected if Z > 1.645 or, equivalently, if the corresponding p-value was less than 0.05.
Time Frame: Peri-procedural
Population: All adverse events reported by the sites were independently adjudicated by the data safety monitory, DSM.
Measure: Number; unit: Pulmonary Veins
Units Other Than Participants: Pulmonary Veins
Arm/Group | Manual Lasso Navigation | Vdrive Lasso Navigation
Number analyzed (Participants) | 43 | 77
Number analyzed (Pulmonary Veins) | 167 | 301
Pulmonary Veins | 167 | 295
Statistical Analysis 1: Comparison: Manual Lasso Navigation vs Vdrive Lasso Navigation; The primary effectiveness endpoint is the successful navigation and EGM recording of each pre-specified pulmonary vein (PV). The RF ablation treatment was not part of the investigational procedure. The null hypothesis was to be tested at the α = 0.05 significance level using a test statistic Z based on the Farrington and Manning likelihood score statistic with adjustment to take into account the correlation between multiple observations (PVs) on the same subject; Test type: Non-Inferiority or Equivalence — The non-inferiority margin d = -0.05. The null hypothesis was to be rejected if Z > 1.645 or, equivalently, if the corresponding p-value was less than 0.05; p = 0.0405, Farrington and Manning — Adjusted to take into account the correlation between multiple PVs on the same subject. The sample estimate of the intraclass correlation coefficient was calculated as the Pearson sample correlation coefficient for all pairs of observations

2. Primary Outcome: Safety Outcome to be Assessed by Comparing the Rate of Adjudicated Serious Adverse Events Within 7 Days of the Procedure Between Both the Control and the Investigational Device Groups.
Description: The Vdrive will allow physicians to manipulate compatible circular mapping catheters while maintaining a safety profile that is not inferior to manual circular catheter navigation. The one-sided null hypothesis was to be tested at the α = 0.05 significance level using a standard unpooled asymptotically normal test statistic. The null hypothesis was to be rejected if Z < -1.7046 or, equivalently, if the corresponding p-value was less than 0.05.
Time Frame: 7 days Follow-up
Measure: Number; unit: participants
Arm/Group | Manual Lasso Navigation | Vdrive Lasso Navigation
Number analyzed (Participants) | 43 | 77
participants | 1 | 3
Statistical Analysis 1: Comparison: Manual Lasso Navigation vs Vdrive Lasso Navigation; Test type: Non-Inferiority or Equivalence — The non-inferiority margin d= 0.07. The one-sided null hypothesis was to be tested at the α = 0.05 significance level using a standard unpooled asymptotically normal test statistic. The null hypothesis was to be rejected if Z < -1.7046 or, equivalently, if the corresponding p-value was less than 0.05; p = .0441, Z-statistic

ADVERSE EVENTS:
Time Frame: If an event was reported by a site as a serious adverse event, SAE, and possibly, probably, or definitely related to the device or the procedure, it is included in the tabulation and the analysis of major adverse events through seven (7) day follow-up.
Description: All adverse events reported by the sites were independently adjudicated by a Data Safety Monitor, DSM.
Arm/Group | Manual Lasso Navigation | Vdrive Lasso Navigation
Serious Adverse Events (participants affected / at risk) | 1/43 | 3/77
Other Adverse Events (participants affected / at risk) | 2/43 | 6/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Manual Lasso Navigation (N=43) | Vdrive Lasso Navigation (N=77)
Pseudoaneurysm (Surgical and medical procedures) | 0 | 1
Cardiac Tamponade (Surgical and medical procedures) | 0 | 1
Bleeding (Surgical and medical procedures) | 0 | 1
Dementia (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Manual Lasso Navigation (N=43) | Vdrive Lasso Navigation (N=77)
Atrial Flutter (Cardiac disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 4
Hematoma (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days